CLINICAL TRIAL: NCT05796388
Title: A Pilot Study to Evaluate the Efficacy and Safety of Virtual Reality in Combination With Linaclotide for the Treatment of Adults With IBS and Constipation Predominance
Brief Title: A Study of Virtual Reality and Linaclotide for IBS-C
Acronym: IBSC-VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Cedars-Sinai Medical Center (Other); AbbVie (Industry); Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Brian Lacy, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-001316
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Virtual reality; IBS-C

STUDY DESIGN:
Intervention Model Description: There will be two groups. One will receive the sham VR the other will receive immersive VR.
Who Masked: Participant, Care Provider
Masking Description: The participant or their treating provider will not know if they have been assigned to the sham VR or immersive VR program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham VR (Sham Comparator): Patients in the sham Virtual Reality group will receive the same brand of head mounted device (Oculus Quest 2), but will only have access to sham content. Both groups will receive standard of care linaclotide treatment 290 mcg.
  Interventions: Device: Virtual Reality
- Immersive VR (Active Comparator): Patients in the immersive Virtual Reality group will receive a head mounted VR device Oculus Quest 2, and will receive active immersive content. Both groups will receive standard of care linaclotide treatment 290 mcg.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Both groups will receive standard of care linaclotide 290 mcg.
  Other Names: Linaclotide

SUMMARY:
The purpose of this study is to determine if adult patients with IBS-C will report an overall greater improvement in IBS symptoms and quality of life when treated with a combination of linaclotide (standard of care medication) and immersive virtual reality (VR) therapy compared to those treated with linaclotide and sham (placebo) VR therapy.

DETAILED DESCRIPTION:
The primary aim of this study will be to assess the benefits of disease-targeted VR combined with linaclotide, compared to sham VR combined with linaclotide, in patients with IBS-C as defined by Rome IV criteria. The investigators hypothesize that compared to patients receiving sham VR and linaclotide, IBS-C patients receiving combination therapy with active VR and linaclotide will achieve statistically significant and clinically meaningful improvements in disease-targeted health-related quality of life while demonstrating improvements in global IBS symptoms, including abdominal pain.

Aims

1. Evaluate changes in quality of life using the validated IBS-QoL (primary outcome);
2. Evaluate global improvement in IBS symptoms using the validated IBS-SSS;
3. Assess global improvement in IBS symptoms using the validated Abdominal Scoring system (11);
4. Evaluate improvement in abdominal pain using a numerical rating system (NRS);
5. Assess improvement in constipation using the Bristol Stool Form Scale (BSFS);
6. Evaluate response to bloating using the validated Mayo bloating questionnaire (12);
7. Assess response to coexisting psychological distress using the validated HADs questionnaire;
8. Evaluate changes in work productivity using the validated WPAI.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (18-70) who meet Rome IV criteria for IBS-C.
* Patients will be required to score below 65 points on the IBS Quality of Life (IBS-QOL) instrument, indicating a score consistent with at least moderate HRQOL (Health-related quality of life) impairment.

Exclusion Criteria:

* Patients will be excluded from the study if they have a comorbid disorder that may confound the diagnosis of IBS, including celiac disease, inflammatory bowel disease, autoimmune disorders that affect the GI system, history of bowel resection, HIV/AIDS, diabetes with HgA1c >7.0, neuroendocrine tumors, microscopic colitis, lactase deficiency, eosinophilic bowel disease, acute intermittent porphyria, or any other condition that a licensed physician believes can mimic IBS symptoms and undermine diagnostic certitude.
* Patients with severe depression, defined as a score equal to or greater than two standard deviations (SDs) on the NIH PROMIS depression scale, or those with suicidal ideations, will also be excluded and provided with standard resources to support their mental health and referred back to their primary care provider, a member of the study team will follow up with the PCP to ensure the communication was received.
* Patients using regular doses of opioid medications will also be excluded given the often-severe impact of opioids on GI motility and potential for pharmacological visceral hyperalgesia.
* Patients will also be excluded from the study if they do not meet Rome IV criteria for IBS-C,
* have a known seizure disorder,
* if symptoms are thought to represent an organic disorder,
* if they have had prior surgery to the colon,
* if symptoms represent a known pelvic floor disorder,
* if the patient is abusing alcohol,
* or if the patient cannot actively participate in the study for any other reason (e.g., inability to understand English as the VR program is in English only).
* Patients previously treated with linaclotide who reported side effects,
* those currently on linaclotide (any dose),
* and those who did not note an improvement in IBS-C symptoms in the past while on linaclotide will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in IBS symptoms | End of study week 8 compared to baseline
  Measure global changes in IBS symptoms using the validated IBS severity scoring system (IBS-SSS) at week 8 compared to baseline, for patients treated with a combination of linaclotide and immersive VR and compare to those treated with linaclotide and sham VR therapy. IBS-SSS is a composite score of abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life (QoL). Each measure is rated from 0 to 100, with total scores ranging from 0 to 500. < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS.

SECONDARY OUTCOMES:
Measure change in quality of life, using the validated IBS-QoL | Week 8
  Irritable Bowel Syndrome-Quality of Life Measure (IBS-QOL) The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Measure changes in abdominal pain using the NRS | Week 8
  The Abdominal Pain Numeric Rating Scale (NRS) patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Measure changes in bloating using the Mayo bloating questionnaire | week 8
  A 40-item questionnaire to understand the daily impact of symptoms of bloating and distension
Measure changes in psychological distress using the HADs questionnaire; | week 8
  The Hospital Anxiety and Depression Scale (HADs) consists of 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represents 'borderline' and 0-7 'normal'
Measure changes in work productivity using the validated WPAI. | Week 8
  The Work Productivity and Activity Impairment (WPAI) questionnaire consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities

CONTACTS AND LOCATIONS:
Overall Officials: Brain Lacy, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials